CLINICAL TRIAL: NCT04304599
Title: Evaluation of a New Female Urinary Catheter Used for Intermittent Catheterization
Brief Title: Evaluation of a New Female Urinary Intermittent Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOF-0035
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Female Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LoFric Elle (Experimental): New hydrophilic female urinary catheter for single use. Ready-to-Use.
  Interventions: Device: LoFric Elle

INTERVENTIONS:
Device: LoFric Elle — The study device is commercially available (CE-marked). It is a device for female intermittent catheterization. Treatment Period will last for 2 weeks. The angulated handle available with the device must be used by each subject at least 10 times.

SUMMARY:
A prospective, multi-centre, interventional study. All subjects will use the study device for two weeks and the angulated handle available with the device must be used by each subject at least 10 times.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent.
* Females aged 18 years and over.
* Maintained urethra sensibility as judged by the subject. (Can you feel the catheter during catheterization? Yes.).
* Practice intermittent catheterization at least 2 times daily.
* Use catheter size available in the study
* Experienced practitioners of intermittent catheterization defined as a minimum of three months on therapy, but not more than approximately 5 years on therapy.
* Adults able to read, write and understand information given to them regarding the study.

Exclusion Criteria:

* Ongoing, symptomatic UTI at enrolment as judged by investigator. The definition of UTI, is a positive urine culture of ≥10^3 CFU/ml of ≥1 bacterial species and presence of symptoms or signs compatible with UTI with no other identified source of infection.
* Known urethral stricture which, in the opinion of the investigator, could influence the subject's evaluation of the catheters.
* Involvement in the planning and conduct of the study (applies to both Wellspect staff and staff at the study site).
* Previous enrolment in the present study.
* Simultaneous participation in another clinical study that may impact the primary endpoint
* Expected or severe non-compliance to protocol as judged by the investigator and/or Wellspect.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the subjects' Quality of Life when practicing IC using LoFric Elle catheters. | 2 weeks
  Primary objective variable is measured by the Intermittent Self-Catheterization Questionnaire (ISC-Q) total score.

SECONDARY OUTCOMES:
Compliance when practicing IC with LoFric Elle. | 2 weeks
  Used study catheter entire study period with the handle at least 10 times: Y/N.
Satisfaction when practicing IC with LoFric Elle. | 2 weeks
  PRO variables (Wellspect questionnaire).
Versatility as in use of the angulated handle when practicing IC with LoFric Elle. | 2 weeks
  PRO variables (Wellspect questionnaire).
Perception when practicing IC with LoFric Elle. | 2 weeks
  PRO variables (Wellspect questionnaire).
The catheter is perceived as slim and discreet which makes it easy to bring, store, and dispose of without obviously being a catheter. | 2 weeks
  ISC-Q domains convenience and discreetness.
The catheter with or without the angulated handle has an ergonomic design which makes it easy to use. | 2 weeks
  ISC-Q domain ease of use.
The catheter is perceived as ready to use. | 2 weeks
  ISC-Q question 1; it is easy to prepare my catheter for use each time I need it.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Sundqvist, MD, PhD, Principal Investigator — Örebro University Hospital, Sweden; Kaj Stenlöf, Dr., Principal Investigator — Carlanderska Hospital
Locations (4):
- Spain (2):
  - Alicante University General Dr. Balmis Hospital, Alicante
  - Hospital Clinic Barcelona, Barcelona
- Sweden (2):
  - Carlanderska Hospital, Gothenburg
  - Urologiska kliniken, mottagning Universitetssjukhuset Örebro, Örebro, Örebro County